CLINICAL TRIAL: NCT03613506
Title: The Role of TGF-β in Abdominal Radiation Injury and Taking Medicine to Block TGF-β for Protecting Normal Organization
Brief Title: The Role and Intervention of TGF-β in Abdominal Radiation Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Director , Director of radiotherapy and chemotherapy for gastrointestinal tumors,Clinical Professor., Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HBCCS AB-01
Record Dates: First submitted 2018-07-23; First posted 2018-08-03 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Radiotherapy Side Effect; Taking Captopril
MeSH Terms: conditions — Radiation Injuries | interventions — Captopril

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peripheral blood TGF-β content before and after radiotherapy (Experimental)
  Interventions: Drug: Captopril 12.5 Mg

INTERVENTIONS:
Drug: Captopril 12.5 Mg — Taking captopril 12.5mg b.i.d for two months before radiotherapy.

SUMMARY:
This project aims to investigate the relationship between radiation-induced the relationship between elevated peripheral blood TGFβ and complications of radiotherapy,and to analysis of changes in peripheral blood TGFβ levels after abdominal radiotherapy and its relationship with radiotherapy complications.Simultaneously,Patients who underwent abdominal radiotherapy were given captopril (sustained release) to block TGFβ,Whether it can reduce peripheral blood TGFβ levels and reduce radiotherapy complications,to explore the protective effect of blocking TGFβ secretion on normal tissues after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form for this study has been signed
2. Age 18-70 years old, gender is not limited，Pathological diagnosis of patients with advanced malignant tumors，Radiotherapy indications；
3. BED (α/β=10)≥50；ECOG score 0-2；Blood routine：WBC≥3.5×109/L,GRAN≥2.0×109/L,Hb≥90g/L，PLT≥100×109/L;
4. Liver function: ALT or AST ≤ 2.5 times the normal high value (ULN)；Bilirubin ≤ 1.5 × ULN, serum APK ≤ 2.5 × ULN;
5. Renal function：Serum creatinine ≤1.5×ULN, and creatinine clearance ≥60ml/min
6. No organ transplant history
7. Women of childbearing age must undergo a urine pregnancy test within 7 days prior to initiation of treatment and the results are negative and not in lactation
8. Male and female patients of childbearing age agreed to adopt a reliable method of contraception before entering the trial and during the study until 30 days after stopping the drug.

Exclusion Criteria:

1. Patients undergoing chemotherapy or targeted therapy at the same time
2. Long-term use of ACEI or ARB drugs for hypertension
3. This radiotherapy site has been treated with radiotherapy；Combined with severe heart disease or major organ failure
4. Have a history of drug abuse or alcohol addiction
5. Combined active infection
6. Combined with severe malnutrition or severe anemia
7. Human immunodeficiency virus (HIV) infection
8. During pregnancy or lactation
9. Those who are unable to tolerate or may be allergic to the drugs used in this study；Persons without civil capacity or limited capacity for civil conduct；
10. Researchers believe that it is not suitable for inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Study the effect of abdominal radiation therapy on peripheral blood TGFβ levels | 12 weeks
  The levels of TGF-β in peripheral blood of patients before and after radiotherapy were compared.
Blocking TGFβ for protective effect on normal tissues | 12 weeks
  Give two groups of patients captopril (sustained release) 12.5mg b.i.d. for two months,comparing their levels of TGF-β in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Jin Peng, Wuhan, Hubei, China